CLINICAL TRIAL: NCT01420731
Title: Phase 4 Study Back Pain and Male Sexual Disfunction
Brief Title: Back Pain and Male Sexual Disfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, gokcen basaranoglu, MD, Bezmialem Vakif University
Other Study IDs: gbms1
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Marriage, Life Event
Keywords: sexual life, back pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Back pain is a common hormonal disorder in men that may affect the phases of male sexual function. The investigators investigated sexual function in male patients with back pain.

A total of 54 men with back pain and 27 age matched voluntary healthy men who served as the as control group were evaluated with a detailed medical and sexual history, including a international erectile function index (IEFI) questionnaire and the Beck Depression Inventory. Serum prolactin, dehydroepiandrosterone sulfate, free testosterone, androstenedione, 17alpha-hydroxyprogesterone, estradiol, free thyroxin and thyrotropin were measured. These variables were compared statistically between the 2 groups.

DETAILED DESCRIPTION:
A total of 54 men with back pain and 27 age matched voluntary healthy men who served as the as control group were evaluated with a detailed medical and sexual history, including a international erectile function index (IEFI) questionnaire and the Beck Depression Inventory. Serum prolactin, dehydroepiandrosterone sulfate, free testosterone, androstenedione, 17alpha-hydroxyprogesterone, estradiol, free thyroxin and thyrotropin were measured. These variables were compared statistically between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Male patient with back pain
* 20 - 45 years old
* Active sexual life

Exclusion Criteria:

* Younger than 20, older than 45 years old

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20-45 years old,male patients with active sexual life
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gökçen Başaranoğlu, MD, Principal Investigator — Beazialem Vakıf University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)